CLINICAL TRIAL: NCT03053843
Title: Randomized Trial of Mediterranean Diet Plus Extravirgin Olive Oil in the Prevention of Recurrent Arrhythmias. The PREDIMAR (PREvención Con DIeta Mediterránea de Arritmias Recurrentes) Trial
Brief Title: Mediterranean Diet Plus Extravirgin Olive Oil in the Prevention of Recurrent Arrhythmias. The PREDIMAR (PREvención Con DIeta Mediterránea de Arritmias Recurrentes) Trial
Acronym: PREDIMAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundación de investigación HM (Other)
Collaborators: University of Navarra (Other); University Hospital Virgen de las Nieves (Other); Hospital General Universitario de Alicante (Other)
Responsible Party: Principal Investigator, Teresa Barrio, MD, PhD, Fundación de investigación HM
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MeDiet+EVOO after AF ablation
Record Dates: First submitted 2017-02-06; First posted 2017-02-15 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Atrial Fibrillation; Atrial Arrhythmia
Keywords: Atrial fibrillation; Mediterranean Diet; Extra Virgin Olive Oil; Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean diet plus extra virgin olive oil (Experimental): These patients will receive 1 liter of EVOO per week free of charge and dietary advice on how to follow a Mediterranean diet with contacts every two months.
  Interventions: Dietary Supplement: Mediterranean diet plus extra virgin olive oil
- no specific diet (No Intervention): The control group will be assigned to the usual care and patients assigned to this group will not receive any special intervention to follow a particular diet, as occurs in the current clinical practice.

INTERVENTIONS:
Dietary Supplement: Mediterranean diet plus extra virgin olive oil — The patients in the intervention group will receive 1 liter of EVOO per week free of charge and dietary advice on how to follow a Mediterranean diet with contacts every two months. Dietary intervention will be carried out by nutritionists with previous experience in the PREDIMED study. All of them were registered, trained and certified for developing the PREDIMED intervention protocol that is similar to the one to be carried out in this study. The theoretical sessions with patients about dietary education shall be conducted in telephone form, using the internet and sending comprehensive written material to their homes that includes recipes, shopping lists, menus and explanations of typical food in the Mediterranean diet
  Arms: Mediterranean diet plus extra virgin olive oil

SUMMARY:
Background: Atrial fibrillation (AF) is the most frequent cardiac arrhythmia and represents a high priority public health problem, as in a few decades it will become a possibly unsustainable load for the national health system. Preventive and therapeutic strategies based on the best possible scientific evidence are required. Ablation therapy, despite being the most effective approach, is associated with a 30-35% arrhythmic recurrence rate. An intervention with Mediterranean diet and extra virgin olive oil (EVOO) has proven effective in primary prevention and reduced the incidence of AF in high-risk subjects in a recent, large, randomized trial (PREDIMED).

Methods: Parallel, randomized, multicenter nutritional intervention trial in 640 patients with AF treated with catheter ablation. Two groups will be randomized in a 1:1 ratio: 1) intervention with Mediterranean diet and EVOO; 2) usual care (control group). The primary objective will be the incidence of atrial tachyarrhythmias for two years after ablation. At least 190 recurrences are expected after 2 years (median) of follow-up. A relative risk of 0.7 is assumed and statistical power of 80%. Follow-up visits will be scheduled at 3, 6, 12, 18 and 24 months. In addition to the in-person visits, event monitors will be used to document episodes. Dietary intervention will be carried out by nutritionists who will use methods adapted from the PREDIMED trial with contacts every 2 months. 1 liter of EVOO per week will be provided for free in the intervention arm. Inflammatory markers will be analyzed in both groups during follow-up. Cox models will be used to estimate adjusted hazard ratios.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic paroxysmal AF (with evidence of more than one symptomatic episode in the last year and at least one documented episode) upon whom catheter ablation is performed.
* Patients with persistent symptomatic AF upon whom catheter ablation is performed.

Exclusion Criteria:

* Serious medical condition that prevents dietary intervention (gastrointestinal disease with intolerance to fats, advanced malignancy, neurological, psychiatric or severe endocrine disease)
* Any other pathology or medical condition that limits survival to less than one year; Immunodeficiency or HIV-positive,
* Consumption of illegal drugs,
* Chronic alcoholism or total consumption of alcohol >80 g/d
* Body mass index > 40 kg/m 2,
* Difficulty or major inconvenience with changing dietary habits, inability to follow a style of Mediterranean diet, low probability of changing dietary habits according to the models of Prochaska and Diciemente (Nigg, 1999)
* History of food allergy or hypersensitivity to any component of EVOO
* Participation in a clinical trial carried out with drugs or use of a drug in experimental state during the year prior to inclusion
* Institutionalized patients for chronic treatment, with lack of autonomy and with inability to perform the clinical follow-up,
* Impossibility of telephone contact
* Patients with acute infection or inflammatory process (e.g. pneumonia) may be included in the study three months after the resolution of the infectious symptoms.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
atrial tachyarrhythmias documented by electrocardiogram or recorder device | mean follow up of 2 years
  Atrial tachyarrhythmia is defined at any fast rate (>100 bpm) of supraventricular origin lasting more than 30 seconds and that is documented by ECG, Holter or event monitor.

SECONDARY OUTCOMES:
Atrial fibrillation documented by electrocardiogram or recorder device | mean follow up of 2 years
  AF is defined at any irregular atrial rhythm lasting more than 30 seconds and that is documented by ECG, Holter or event monitor. AF may or may not be symptomatic.
changes in Inflammatory markers in blood samples | 1 year follow up
  Prior to ablation blood samples will be collected for determination of inflammatory parameters in a subsample of the study (neutrophil to lymphocyte ratio, TNF-alpha, fibrinogen, IL-2, IL6, IL-8, C-reactive protein). At 3 and 12 months of follow-up the determination of these parameters will be repeated.
Changes in quality of life measured by SF-36 questionnaire | mean follow up of 2 years
  Change in quality of life during the follow up measured by SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Martinez González, MD, PhD, MPH, Study Chair — University of Navarra; Jesus Almendral Garrote, MD, PhD, FESC, Study Director — Fundación HM; Teresa Barrio Lopez, MD, PhD, Principal Investigator — Fundación HM
Locations (2):
- Spain (2):
  - Teresa Barrio Lopez, Madrid
  - Teresa Barrio López, Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Martinez-Gonzalez MA, Toledo E, Aros F, Fiol M, Corella D, Salas-Salvado J, Ros E, Covas MI, Fernandez-Crehuet J, Lapetra J, Munoz MA, Fito M, Serra-Majem L, Pinto X, Lamuela-Raventos RM, Sorli JV, Babio N, Buil-Cosiales P, Ruiz-Gutierrez V, Estruch R, Alonso A; PREDIMED Investigators. Extravirgin olive oil consumption reduces risk of atrial fibrillation: the PREDIMED (Prevencion con Dieta Mediterranea) trial. Circulation. 2014 Jul 1;130(1):18-26. doi: 10.1161/CIRCULATIONAHA.113.006921. Epub 2014 Apr 30. PMID 24787471
- [Result] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary prevention of cardiovascular disease with a Mediterranean diet. N Engl J Med. 2013 Apr 4;368(14):1279-90. doi: 10.1056/NEJMoa1200303. Epub 2013 Feb 25. PMID 23432189 (Retraction: PMID 29897867 N Engl J Med. 2018 Jun 21;378(25):2441-2442)
- [Derived] Goni L, de la O V, Barrio-Lopez MT, Ramos P, Tercedor L, Ibanez-Criado JL, Castellanos E, Ibanez Criado A, Macias Ruiz R, Garcia-Bolao I, Almendral J, Martinez-Gonzalez MA, Ruiz-Canela M. A Remote Nutritional Intervention to Change the Dietary Habits of Patients Undergoing Ablation of Atrial Fibrillation: Randomized Controlled Trial. J Med Internet Res. 2020 Dec 7;22(12):e21436. doi: 10.2196/21436. PMID 33284131
- [Derived] Barrio-Lopez MT, Ruiz-Canela M, Ramos P, Tercedor L, Ibanez Criado JL, Ortiz M, Goni L, Ibanez Criado A, Macias-Ruiz R, Garcia-Bolao I, Martinez-Gonzalez MA, Almendral J. PREvention of recurrent arrhythmias with Mediterranean diet (PREDIMAR) study in patients with atrial fibrillation: Rationale, design and methods. Am Heart J. 2020 Feb;220:127-136. doi: 10.1016/j.ahj.2019.10.009. Epub 2019 Oct 26. PMID 31809992